CLINICAL TRIAL: NCT05587413
Title: Effectiveness of Periodontal Treatment for the Glycemic Conttrol of Type II Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Gul Muhammad Shaikh, Doctor, University of Lahore
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: UIPH/UOL/193/2019
Record Dates: First submitted 2022-10-12; First posted 2022-10-20 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental)
  Interventions: Procedure: periodontal care
- control group (No Intervention)

INTERVENTIONS:
Procedure: periodontal care — periodontal treatment
  Arms: treatment group

SUMMARY:
The project is intended to find out the effect of Periodontal treatment for the glycemic control of type II diabetes mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having Diabetes Mellitus and diagnosed with Periodontitis for last six months.
2. Aged between 30-60 years.
3. Patients with HbA1C level 7-9.5%, measured within three months prior to present study.

Exclusion Criteria:

1. Patients with acute oral infection
2. Need for immediate tooth extractions
3. Severe Hypertension (>180/110 mm Hg)
4. Edentulous Patients
5. Patients with Diabetic Nephropathy
6. Patients with Diabetic Retinopathy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-11-02 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1C between the control group and interventional group. | one year
  The primary outcome of the trial

CONTACTS AND LOCATIONS:
Locations (1):
- Uol, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
will be informed